CLINICAL TRIAL: NCT03763305
Title: Comparison of Skin Sympathetic Nerve Activity According to Different Anesthetics During Transurethral Procedures
Brief Title: Comparison of Skin Sympathetic Nerve Activity According to Different Anesthetics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices for measuring SKNA are need to be re-constructed, which takes considerable time.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SKNA-TURB
Record Dates: First submitted 2018-11-25; First posted 2018-12-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: SKNA According to Different Anesthetics
Keywords: skin sympathetic nerve activity, anesthetics
MeSH Terms: interventions — Propofol; Remifentanil; Sevoflurane; Desflurane; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total intravenous anesthesia (TIVA) (Experimental): Study participants are anesthetized by total intravenous anesthesia (TIVA) using propofol continuous infusion and remifentanil continuous infusion. During induction of general anesthesia, participants receive 3~5mcg/mL Propofol Fresenius and 3~5ng/mL and Remifentanil [Ultiva] as initial effect site concentrations. The effect site concentration is controlled with target-controlled infusion to maintain bispectral index (BIS) values between 40 and 60.
  Interventions: Drug: Propofol continuous infusion; Drug: Remifentanil
- Sevoflurane (Experimental): Study participants receive fentanyl 1mcg/kg and propofol bolus injection 1.5~2mg/kg for induction of general anesthesia. For maintenance of anesthesia, sevoflurane inhalant solution [Sojourn] is used to maintain 1 age-related minimum alveolar concentration (MAC).
  Interventions: Drug: Sevoflurane; Drug: Propofol bolus injection; Drug: Fentanyl
- Desflurane (Experimental): Study participants receive fentanyl 1mcg/kg and propofol bolus injection 1.5~2mg/kg for induction of general anesthesia. For maintenance of anesthesia, desflurane [Suprane] is used to maintain 1 age-related minimum alveolar concentration (MAC).
  Interventions: Drug: Desflurane; Drug: Propofol bolus injection; Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol continuous infusion — Propofol intravenous continuous infusion for anesthetic induction and maintenance
  Other Names: Propofol Fresenius
  Arms: Total intravenous anesthesia (TIVA)
Drug: Remifentanil — Remifentanil intravenous continuous infusion for anesthetic induction and maintenance
  Other Names: Ultiva
  Arms: Total intravenous anesthesia (TIVA)
Drug: Sevoflurane — Study participants receive fentanyl 1mcg/kg and propofol 1.5~2mg/kg for induction of general anesthesia. For maintenance of anesthesia, desflurane is used to maintain 1 age-related minimum alveolar concentration (MAC).
  Other Names: Sevoflurane Inhalant Solution [Sojourn]
  Arms: Sevoflurane
Drug: Desflurane — 1 age-related minimum alveolar concentration (MAC) of desflurane inhalation for anesthetic maintenance
  Other Names: Desflurane Inhalation Solution [Suprane]
  Arms: Desflurane
Drug: Propofol bolus injection — Propofol intravenous injection for anesthetic induction
  Other Names: Anepol; Pofol
  Arms: Desflurane; Sevoflurane
Drug: Fentanyl — Fentanyl intravenous injection for anesthetic induction
  Arms: Desflurane; Sevoflurane

SUMMARY:
Skin sympathetic nerve activity (SKNA) has recently been discovered from the electrocardiogram obtained from healthy volunteers. The raw physiologic electric signal from electrodes placed on the skin was reprocessed through filtering and integration using software to produce the SKNA signal. However, no study has yet provided knowledge on the effect of anesthetics on SKNA during general anesthesia.

DETAILED DESCRIPTION:
The most commonly used anesthetic techniques during general anesthesia are the total intravenous anesthesia (TIVA) and anesthesia using inhalants such as sevoflurane or desflurane. For TIVA, the combination of propofol and remifentanil has been used and remifentanil is known for increasing vagal tone and inhibiting sympathetic nervous system as other opioids do. Sevoflurane is presumed to have no effect on parasympathetic or sympathetic tone. On the other hand, desflurane induces tachycardia and is noted for activating sympathetic activity. Previous studies on sympathetic nervous activity according to different anesthetics did not directly measure sympathetic tone but have relied on indirect measures such as blood pressure, heart rate, and heart rate variability.

In order to evaluate skin sympathetic nerve activity according to different anesthetics, we will be recruiting patients undergoing transurethral procedures, where the sympathetic tone is expected to be activated during anesthesia and surgery. The transurethral procedures consist of transurethral resection of bladder (TURB) and transurethral resection of prostate (TURP). During transurethral surgery, about 300mL of fluid is used to fill the bladder to secure surgical view and for irrigation. Bladder expansion causes sympathetic nerve activation and vasoconstriction, which will also increase SKNA signals. The purpose of this study is to measure skin sympathetic nerve activity according to different anesthetics during intraoperative events that stimulate sympathetic tone.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective transurethral procedures under general anesthesia

Exclusion Criteria:

* Diagnosed with autonomic dysfunction
* Current use of beta blockers
* Cardiac arrhythmia
* Absolute indication for either TIVA or inhalants, absolute contraindication for either TIVA or inhalants (adverse effects on either propofol or remifentanil, risk of malignant hyperthermia)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The skin sympathetic nerve activity (SKNA) presented as uV obtained via skin leads. | Intraoperative
  The average intraoperative SKNA divided by average SKNA before induction of general anesthesia (T0)

SECONDARY OUTCOMES:
Percent change of SKNA | T1: 1.5 minute after use of anesthetics, T2: 1.5 minute after use of muscle relaxant, T3: 30 seconds after intubation, T4: before bladder expansion, T5: 30 seconds after bladder expansion, T6: 30 sec after start of surgery, T7: 30sec after end of surgery
  Percent change of SKNA at different time points (T1-T7) compared to T0

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Study Director — Seoul National University Hospital